CLINICAL TRIAL: NCT04385082
Title: Sex-dependent Effects of Cannabis: Assessing Analgesic, Abuse-related and Pharmacokinetic Differences Between Men and Women
Brief Title: Cannabis Effects as a Function of Sex
Acronym: CanSex
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: University of California, Los Angeles (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Principal Investigator, Ziva D. Cooper, PhD, Associate Professor, University of California, Los Angeles
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: 19-000876; R01DA047296 (NIH)
Record Dates: First submitted 2020-05-07; First posted 2020-05-12 (Actual); Last update posted 2025-05-13 (Actual); Status verified 2025-05

CONDITIONS: Pain; Abuse, Drug
Keywords: Pain; Cannabis; THC
MeSH Terms: conditions — Pain; Substance-Related Disorders; Marijuana Abuse

STUDY DESIGN:
Intervention Model Description: This is a randomized, double-blind, placebo-controlled study. All participants will complete all dose conditions in a randomized order.
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- Placebo (Placebo Comparator): Smoked Cannabis (~0% THC)
  Interventions: Drug: Placebo Cannabis
- Low strength cannabis (Experimental): Smoked Cannabis (~4% THC)
  Interventions: Drug: Active Cannabis
- Higher strength cannabis (Experimental): Smoked Cannabis (~10% THC)
  Interventions: Drug: Active Cannabis

INTERVENTIONS:
Drug: Active Cannabis — Smoked cannabis with THC
  Arms: Higher strength cannabis; Low strength cannabis
Drug: Placebo Cannabis — Placebo smoked cannabis (no THC)
  Arms: Placebo

SUMMARY:
The purpose of this research is to assess the impact of cannabis on the analgesic and abuse-related effects between men and women

DETAILED DESCRIPTION:
The proposed study will compare smoked cannabis's dose-dependent, analgesic and abuse-related effects between men and women and variables that underlie these sex-dependent differences, including pharmacokinetics of THC.

ELIGIBILITY:
Inclusion Criteria:

* Male or non-pregnant female aged 21-55 years
* Report use of cannabis an average of 1-7 days per week
* Not currently seeking treatment for their cannabis use
* Urine test positive for recent cannabis use for heavy users
* No reported adverse effects with cannabis smoking in light users
* Have a Body Mass Index from 18.5 - 34kg/m2.
* Able to perform all study procedures
* FEMALES: Currently practicing a non-hormonal effective form of birth control
* FEMALES: Must be regularly cycling

Exclusion Criteria:

* Meeting DSM-V criteria for any substance use disorder other than nicotine, caffeine, or cannabis use disorder
* Report using other illicit drugs in the prior 4 weeks
* History or current evidence of severe psychiatric illness or medical condition judged by the study physician and PI to put the participant at greater risk of experiencing adverse events due to completion of study procedures, interfere with their ability to participate in the study, or their capacity to provide informed consent.
* Current use of medical cannabis, prescription analgesics, or any medications that may affect study outcomes
* Current pain
* Insensitivity to the cold water stimulus of the Cold Pressor Test
* FEMALES: using a hormonal contraceptive

Ages: 21 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 160 (Estimated)
Dates: Start 2021-07-08 (Actual); Primary Completion 2025-12-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Subject-rated drug effects | 5 hours
  Average and peak subjective ratings of drug effects associated with abuse liability as measured using visual analogue scales (VAS; 1-100mm).
Analgesia as measured using the Cold Pressor Test | 5 hours
  Peak and average pain threshold and tolerance assessed using the Cold Pressor Test
Pharmacokinetics of THC and metabolites | 5 hours
  Plasma levels of THC, 11-OH-THC, and THCCOOH

SECONDARY OUTCOMES:
Drug reinforcement using the cannabis self-administration task | 5 hours
  Average number of cannabis puffs self-administered as a function of cannabis strength and sex. For this task, up to three 'puffs' of cannabis may be chosen for self-administration during each session.

CONTACTS AND LOCATIONS:
Overall Officials: Ziva Cooper, PhD, Principal Investigator — University of California, Los Angeles
Locations (1):
- University of California, Los Angeles, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: No